CLINICAL TRIAL: NCT02335125
Title: A Policy Relevant US Trauma Care System Pragmatic Trial for PTSD and Comorbidity Pilot
Acronym: TSOS6
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Douglas Zatzick, Professor, Psychiatry & Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00010782; UH2MH106338 (NIH)
Record Dates: First submitted 2014-11-14; First posted 2015-01-09 (Estimated); Results first posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Posttraumatic Stress Disorder; Depression; Alcohol-Related Disorders; Suicidal Ideation; Substance-Related Disorders; Mild Cognitive Impairment; Quality of Life
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Alcohol-Related Disorders; Suicidal Ideation; Substance-Related Disorders; Cognitive Dysfunction | interventions — Motivational Interviewing; Psychotropic Drugs

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The intervention aims to prevent the development of chronic PTSD and depressive symptoms, alcohol use problems, and enduring physical disability in survivors of both TBI and non-TBI injuries. The intervention utilizes a computerized decision support tool to flexibly target these multiple conditions including and includes care management, medication, and psychotherapy elements.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Cognitive Behavioral Therapy Elements; Drug: Psychotropic Drugs; Other: Care Management
- Usual Care (No Intervention): Only standard care practices will be administered to this arm.

INTERVENTIONS:
Behavioral: Motivational Interviewing
  Arms: Intervention
Behavioral: Cognitive Behavioral Therapy Elements
  Arms: Intervention
Drug: Psychotropic Drugs
  Arms: Intervention
Other: Care Management
  Arms: Intervention

SUMMARY:
The goal of this pilot study is to develop and implement a larger scale, multi-site stepped collaborative care trial that targets injured patients with presentations of posttraumatic stress disorder (PTSD) and related comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient/Emergency Admission for traumatic injury

Exclusion Criteria:

* Non-English speaking
* Self-inflicted injury
* Actively psychotic
* Incarcerated or in custody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Zatzick, MD, Principal Investigator — University of Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: The intervention aims to prevent the development of chronic PTSD and depressive symptoms, alcohol use problems, and enduring physical disability in survivors of both TBI and non-TBI injuries. The intervention utilizes a computerized decision support tool to flexibly target these multiple conditions including and includes care management, medication, and psychotherapy elements.
  Motivational Interviewing
  Cognitive Behavioral Therapy Elements
  Psychotropic Drugs
  Care Management
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 18 | 13 | 31
  >=65 years | 1 | 5 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (18.1) | 48.4 (18.9) | 46.0 (18.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 14 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 16 | 11 | 27
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline PTSD Checklist Civilian (PCL-C) at 1 Month
Description: The investigators will use the PTSD Checklist - Civilian (PCL-C). The scoring of the scale ranges from a minimum of 17 to a maximum of 85, with higher scores indicating a worse outcome. The measure can also provide a rating of symptoms consistent with a diagnosis of PTSD.
Time Frame: Baseline and 1-month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 20
score on a scale | 1.30 [-4.81 to 7.42] | 5.04 [-1.07 to 11.15]

2. Primary Outcome: Change From Baseline Alcohol Use Disorders Identification at 1 Month
Description: The investigators will use the Alcohol Use Disorders Identification Test (AUDIT) as a continuous measure. The 10-item scale score ranges from 0-40, with higher values indicating a worse outcome.
Time Frame: Baseline and 1-month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 20
score on a scale | -1.36 [-3.38 to 0.66] | -2.31 [-4.38 to -0.25]

3. Primary Outcome: Change From Patient Health Questionnaire 9 Item Depression Scale at 1 Month
Description: The investigators will use the Patient Health Questionnaire 9-item Depression Scale (PHQ-9). The scoring of the scale ranges from a minimum of 0 to a maximum of 27, with higher scores indicating a worse outcome.
Time Frame: Baseline and 1-month
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 20
score on a scale | 1.27 [-1.20 to 3.74] | 0.28 [-2.25 to 2.82]

4. Secondary Outcome: Change in Functional Status
Description: The investigators will use the Medical Outcomes Study Short Form healthy survey (MOS SF-12/36) physical components summary to assess physical function. The minimum and maximum scores are 0-100 with higher scores representing a better outcome.
Time Frame: Baseline and 1-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 48.2 (12.2) | 46.5 (12.1)
  1 Month | 30.1 (13.6) | 33.0 (9.1)

5. Secondary Outcome: Patient Health Questionnaire Item 9 Suicide Question
Description: Item 9 of the Patient Health Questionnaire 9-item (PHQ-9) scale assesses suicidal ideation. It is scored from 0 to 3, with a score of 1 or greater indicating a patient has suicidal ideation. Participants with a PHQ-9 item 9 score of greater than or equal to 1 are reported for this outcome.
Time Frame: Baseline and 1-month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 20
Participants
  Baseline | 3 | 2
  1 Month | 4 | 6

6. Secondary Outcome: Number of Participants Endorsing a Single Item That Assesses Drug Use
Description: Single items that assess drug use across multiple substances (e.g., Cocaine, Prescription Opiates). Single item self-report dichotomized as none versus at least monthly use.
Time Frame: Baseline and 1-month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 20
Participants
  Baseline | 12 | 10
  1 Month | 15 | 13

7. Secondary Outcome: Cognitive Impairment Scale
Description: The investigators will use the National Study on the Costs and Outcomes of Trauma (NSCOT) Cognitive Screen, a 4 - Item Traumatic Brain Injury / Post-concussive Symptom Screen. The scoring of the scale ranges from a minimum of 4 to a maximum of 20, with lower scores indicating a worse outcome.
Time Frame: Baseline and 1-month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 16.3 (3.3) | 16.9 (3.4)
  1 Month | 16.3 (4.1) | 15.9 (4.1)

8. Other Pre Specified Outcome: Chronic Medical Condition ICD-9 Definition
Description: Moderating Variable
Time Frame: Baseline
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Traumatic Brain Injury Status ICD-9 Definition
Description: Moderating Variable
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=20) | Usual Care (N=20)
Surgical complication unrelated to study participation which resulted in death (Surgical and medical procedures) | 1 | 0 — Site 1 recruited a subject on while he was inpatient and completed his baseline interview. Five days later, the subject went in to surgery while still inpatient for repair work on his ankle. The subject died while in surgery.

LIMITATIONS AND CAVEATS:
During the pilot study roll-out it was noted that rather than characterizing trauma center providers as staff versus care managers, that a better characterization was to split staff across two trauma centers; this update was made on 2/6/19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes